CLINICAL TRIAL: NCT01032200
Title: A Feasibility Study of Armodafinil for Brain Radiation-Induced Fatigue
Brief Title: Armodafinil in Treating Fatigue Caused By Radiation Therapy in Patients With Primary Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00012856; U10CA081851 (NIH); REBACCCWFU97509 (Other: NCI)
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Brain Tumors; Nervous System Tumors; Cognition Disorders; Fatigue
Keywords: fatigue; cognitive/functional effects; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult pineal gland astrocytoma; adult subependymal giant cell astrocytoma; adult oligodendroglioma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic meningioma; adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult papillary meningioma; adult brain stem glioma
MeSH Terms: conditions — Brain Neoplasms; Nervous System Neoplasms; Cognition Disorders; Fatigue; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma; Ependymoma; Glioma, Subependymal; Meningioma | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Armodafinil (Experimental): Patients receive oral armodafinil once daily beginning no later than the fifth fraction of brain radiotherapy and continuing for 9-11 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: Armodafinil
- Arm II - Placebo (Placebo Comparator): Patients receive oral placebo once daily beginning no later than the fifth fraction of brain radiotherapy and continuing for 9-11 weeks in the absence of unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Armodafinil — Given orally
  Arms: Arm I - Armodafinil
Other: placebo — Given orally
  Arms: Arm II - Placebo

SUMMARY:
RATIONALE: Armodafinil may help relieve fatigue and improve quality of life in patients with cancer receiving radiation therapy to the brain.

PURPOSE: This clinical trial is studying how well armodafinil works in treating fatigue caused by radiation therapy in patients with primary brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate study accrual, adherence, retention, and participation of patients with primary brain tumors undergoing partial- or whole-brain radiotherapy who are randomized to receive armodafinil or placebo.
* To estimate the variability of fatigue, quality of life, and neurocognitive function in these patients.

Secondary

* To obtain a preliminary estimate of the effect of armodafinil on fatigue as measured by the fatigue subscale of the FACIT-F and the Brief Fatigue Inventory.
* To estimate the rates of toxicity and adverse events associated with armodafinil.
* To obtain preliminary estimates of the effect of armodafinil on sleepiness as measured by the Epworth Sleep Scale; overall quality of life and brain-specific quality of life as measured by the FACT-G with the brain subscale; and cognitive function as measured by a comprehensive Wake Forest Cognitive Function Battery.

OUTLINE: This is a multicenter study. Patients are stratified according to therapy (radiotherapy alone vs radiotherapy and chemotherapy) and Karnofsky performance status (60-80% vs 90-100%). Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral armodafinil once daily beginning no later than the fifth fraction of brain radiotherapy and continuing for 9-11 weeks in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily beginning no later than the fifth fraction of brain radiotherapy and continuing for 9-11 weeks in the absence of unacceptable toxicity.

Patients complete questionnaires assessing fatigue, quality of life, and neurocognitive function at baseline and periodically during study.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed primary brain tumor, including any of the following:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Low-grade glioma
  * Meningioma
  * Ependymoma
  * Other primary brain tumor histologies
* Planning to undergo external-beam cranial radiotherapy (partial- or whole-brain radiotherapy) meeting all of the following criteria:

  * Total dose ≥ 4,500 cGy
  * Total number of fractions ≥ 25 fractions
  * Dose per fraction ≥ 150 cGy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Hemoglobin ≥ 10.0 g/dL (erythropoietin or transfusion allowed for symptomatically anemic patients with a hemoglobin < 10 g/dL)
* Creatinine ≤ 2 mg/dL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Sexually active women of childbearing potential must use a reliable method of birth control

  * It is recommended that patients use non-hormonal contraceptives, in addition to or in place of hormonal contraceptives, during and for one month following treatment with armodafinil
* Prior malignancies allowed

Exclusion Criteria:

* No baseline headaches (i.e., headaches occurring in the week before baseline assessment) of grade 4 severity (defined as severe and disabling headaches, requiring analgesics, and interfering with and preventing function or activities of daily living)
* No concurrent uncontrolled illness that may cause fatigue; interfere with drug absorption, distribution, metabolism, or excretion; or limit compliance with study requirements including, but not limited to, any of the following:

  * Ongoing or active infection
  * Chronic renal insufficiency
  * Psychiatric illness (psychosis, psychotic disorder, history of suicide attempt, or actively suicidal)
  * Extreme social situations (e.g., transportation issues that would preclude study compliance)
* Patients with a history of cardiac issues (symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia) should not use armodafinil as it may cause chest pain, palpitations, dyspnea, and transient ischemic T-wave changes on ECG
* No history of allergic reaction attributed to modafinil or armodafinil
* No anticipated or planned excessive consumption of coffee, tea, and/or caffeine-containing beverages averaging > 600 mg of caffeine/day (i.e., approximately 6 cups of coffee/day, 12 cups of hot tea/day, or 12 cans of cola/day)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior fractionated external-beam cranial radiotherapy
* More than 30 days since prior monoamine oxidate inhibitors or investigational drugs
* More than 2 weeks since prior and no concurrent modafinil (Provigil), donepezil (Aricept), memantine hydrochloride (Namenda), methylphenidate (Ritalin), dextroamphetamine-amphetamine (Adderall), ginkgo biloba, or any other cognitive function-enhancing drugs
* At least 4 weeks since prior and no concurrent interstitial or intracavitary chemotherapy and/or radiotherapy or stereotactic radiosurgery (i.e., Gamma Knife, Linac, or Cyberknife)
* No concurrent erythropoietin, transfusion, or iron therapy (unless patient is symptomatically anemic with hemoglobin < 10 g/dL)
* Concurrent chemotherapy allowed
* Concurrent hormonal therapy for other malignancies allowed

  * No concurrent non-hormonal therapy (e.g., Herceptin and other targeted agents), or cytotoxic chemotherapy
* No concurrent clopidogrel bisulfate (Plavix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2013-01-08 (Actual); Study Completion 2013-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
Started | 26 | 28
Completed | 22 | 21
Not Completed | 4 | 7
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Toxicity | 0 | 2
Not completed — Progression | 1 | 0
Not completed — Multiple | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Armodafinil | Arm II - Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 7 | 10 | 17
Age, Continuous [Median (Full Range); unit: years] | 59 [28 to 78] | 58 [29 to 79] | 59 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Retention is defined as the percentage of participants who complete the 4 week post-RT questionnaires.
Time Frame: 4 weeks post-RT (approximately 3 months post randomization)
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
Number analyzed (Participants) | 26 | 28
percentage of participants | 85 | 75

2. Primary Outcome: Adherence
Description: Adherence is the percentage of ideal number of pills taken while on study (based on returned diaries)
Time Frame: 4 weeks post-RT (approximately 3 months post randomization)
Population: Participants who returned pill diaries
Measure: Mean (Full Range); unit: percentage of ideal number of pills
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
Number analyzed (Participants) | 22 | 25
percentage of ideal number of pills | 92.6 [0 to 100] | 95.7 [70.3 to 100]

3. Secondary Outcome: Fatigue
Description: Fatigue is measured by the fatigue subscale of the Functional Assessment of Chronic Illness Therapy Questionnaire. It consists of 13 questions each answered on a 0 to 4 scale. The fatigue score is the sum of the responses with some questions reverse scored. The total Score ranges from 0 to 52, with higher scores indicating less fatigue.
Time Frame: 4 weeks post-RT
Population: Participants with any data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
Number analyzed (Participants) | 26 | 27
units on a scale | 32.4 (2.6) | 36.4 (2.5)

4. Secondary Outcome: Sleepiness
Description: Sleepiness as measured by the Epworth Sleep Scale. It consists of 8 questions that measure daytime sleepiness in which the patient records their likelihood of dozing or sleeping during a number of routine daily activities. ESS scores range from 0 to 24. Higher scores denote greater sleepiness.
Time Frame: 4 weeks post-RT
Population: Participants with any data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
Number analyzed (Participants) | 26 | 27
units on a scale | 7.2 (1.0) | 8.3 (1.0)

5. Secondary Outcome: HVLT-IR
Description: HVLT-IR is the Hopkins Verbal learning test - immediate recall. Participants are given 12 words to remember. They are then asked to recall those words. This is repeated 3 times. Minimum recalled words 0 maximum 36. The HVLT-IR score is the sum of correctly recalled words across the three trials. Higher scores indicate better recall.
Time Frame: 4 weeks post-RT
Population: Participants with any data
Measure: Least Squares Mean (Standard Error); unit: number of correctly recalled words
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
Number analyzed (Participants) | 26 | 27
number of correctly recalled words | 21.2 (1.5) | 20.0 (1.4)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The denominator for adverse events in each arm is the number of participants who provided post-treatment data.
Arm/Group | Arm I - Armodafinil | Arm II - Placebo
All-Cause Mortality (participants affected / at risk) | 1/26 | 2/28
Serious Adverse Events (participants affected / at risk) | 10/26 | 8/27
Other Adverse Events (participants affected / at risk) | 26/26 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Armodafinil (N=26) | Arm II - Placebo (N=27)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Agitation (General disorders) | 0 (0) | 2 (2)
Alanine Aminotransferase Increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anxiety (General disorders) | 1 (1) | 1 (2)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Delirium (General disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1) | 1 (1)
Muscle Weakness - left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Weakness - lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Optic Nerve Disorder (Eye disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Personality Change (Psychiatric disorders) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Armodafinil (N=26) | Arm II - Placebo (N=27)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (11) | 6 (15)
Anxiety (Psychiatric disorders) | 15 (55) | 10 (39)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 7 (18)
Back Pain (General disorders) | 2 (3) | 3 (7)
Blurred Vision (Eye disorders) | 4 (11) | 2 (3)
Cognitive Disturbance (Psychiatric disorders) | 0 (0) | 2 (10)
Confusion (Psychiatric disorders) | 3 (21) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Dizziness (Ear and labyrinth disorders) | 9 (24) | 8 (32)
Dry Mouth (Gastrointestinal disorders) | 9 (32) | 9 (45)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 0 (0)
Ear and Labyrinth - Other (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Edema Limbs (General disorders) | 0 (0) | 2 (2)
Eye Disorders - Other (Eye disorders) | 5 (15) | 0 (0)
Fatigue (General disorders) | 17 (95) | 17 (71)
Gait Disturbance (General disorders) | 0 (0) | 2 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (8)
Headache (General disorders) | 19 (93) | 16 (53)
Hypertension (Cardiac disorders) | 3 (7) | 5 (21)
Insomnia (Psychiatric disorders) | 12 (46) | 14 (63)
Investigations - Other (Investigations) | 0 (0) | 2 (2)
Localized Edema (General disorders) | 2 (12) | 3 (15)
Memory Impairment (Psychiatric disorders) | 0 (0) | 5 (17)
Mucosal Infection (Infections and infestations) | 4 (16) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (35) | 13 (23)
Pain (General disorders) | 3 (10) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (7) | 2 (3)
Rash Masculo-Papular (Skin and subcutaneous tissue disorders) | 7 (15) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 5 (5)
Thromboembolic Event (Vascular disorders) | 3 (6) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (11)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 3 (5)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less